CLINICAL TRIAL: NCT02545088
Title: New Technology for Individualised, Intensive Training of Gait After Stroke- Phase II Trials, Study II
Brief Title: New Technology for Individualised, Intensive Training of Gait After Stroke- Study II
Acronym: HAL-RCT-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danderyd Hospital (Other)
Collaborators: University of Tsukuba (Other); Sahlgrenska University Hospital (Other); Umeå University (Other)
Responsible Party: Principal Investigator, Susanne Palmcrantz, PhD, Reg physiotherapist, Danderyd Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAL-RCT-Phase II-Study II
Record Dates: First submitted 2015-08-24; First posted 2015-09-09 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Stroke; Ambulation Difficulty; Hemiparesis
Keywords: Rehabilitation; Robotics
MeSH Terms: conditions — Stroke; Mobility Limitation; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Study group Hybrid Assistive Limb (HAL) (Experimental)
  Interventions: Device: Hybrid Assistive Limb (HAL)
- 1st control group (Active Comparator)
  Interventions: Other: 1st control group
- 2nd control group (Active Comparator)
  Interventions: Other: 2nd control group

INTERVENTIONS:
Device: Hybrid Assistive Limb (HAL) — Intensive gait training with Hybrid Assistive Limb (HAL) is performed 1 session/day, 3 days/week for 6 weeks and each session will not exceed 60 min of effective walking time with HAL. In addition, each session will include conventional gait training that will not exceed 30 min effective training time.
  Arms: Study group Hybrid Assistive Limb (HAL)
Other: 1st control group — Conventional gait training performed 1 session/day, 3 days/week for 6 weeks that will not exceed 1h 30 min effective training time.
  Arms: 1st control group
Other: 2nd control group — The 2nd control group will not receive an intervention.
  Arms: 2nd control group

SUMMARY:
The overall purpose of this project is to establish the added value of training with the Hybrid Assistive Limb (HAL) exoskeleton system as part of regular rehabilitation intervention programs after stroke.

The main specific aims are:

(i) to compare potential effects on functioning and disability of gait and mobility training long-term after stroke by comparing A) HAL-training combined with conventional rehabilitation interventions to B) conventional rehabilitation interventions without HAL and to C) no intervention.

DETAILED DESCRIPTION:
The effectiveness of the interventions will be assessed in terms aspects of body function, walking ability and endurance as well as level of activity in daily living and participation assessed at the end of intervention and at a 6 and 12 months follow-up.

Intensive gait training with HAL is performed 1 session/day, 3 days/week for 6 weeks and each session will not exceed 60 min of effective walking time with HAL. In addition, each session will include conventional gait training that will not exceed 30 min effective training time. To standardize the training procedure, training with HAL is performed on a treadmill and to enable body weight support. Body weight support is used to prevent falls and to unburden the weight of the suit (9 kg). The training program is performed by physiotherapists, trained in the HAL method and the study procedures. At the end of the 6 weeks, the physiotherapist that has been engaged in the patient's conventional training will perform 1-2 home visits to inform/educate the patient and those who are providing assistance to the patient in how the patient can make use of any gains in gait function during activities of daily living.

The 1st control group will receive conventional gait training performed 1 session/day, 3 days/week for 6 weeks that will not exceed 1h 30 min effective training time.

The 2nd control group will not receive an intervention. The conventional gait training is performed according to current best evidence based practice and may include over ground walking with assistance and/or assistant devices as well as the use of a treadmill and body weight support and training of gait function in activities of daily living

ELIGIBILITY:
Inclusion Criteria:

* 1-10 years since stroke onset
* Able to walk but not independently, i.e. need of manual support or close supervision due to lower extremity paresis, FAC score 2-3 or FAC 4 combined with gait speed <0.8m/s according to 10 meter walk test, which corresponds to limitations in community ambulation (Bowden et al 2008)
* Ability to understand training instructions as well as written and oral study information and to express informed consent or by proxy
* Body size compatible with the HAL suit.

Exclusion Criteria:

* Contracture restricting gait movements at any lower limb joint
* Cardiovascular or other somatic condition incompatible with intensive gait training
* Severe, contagious infections (e.g. Methicillin Resistant Staphylococcus Aureus (MRSA) or Extended Spectrum Beta Lactamase bacteria).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Change in 6 min walk test | Assessment at baseline, after 6 weeks of intervention, 6 and 12 month post intervention
  walking ability and endurance

SECONDARY OUTCOMES:
Fugl Meyer Scale for lower extremities | Assessment at baseline, after 6 weeks of intervention, 6 and 12 month post intervention
  Sensory and motor function in lower extremities
Modified Ashworth Scale | Assessment at baseline, after 6 weeks of intervention, 6 and 12 month post intervention
  Spasticity
Spasticity measured with Neuroflexor foot module | Assessment at baseline, after 6 weeks of intervention, 6 and 12 month post intervention
  Spasticity
Berg Balance Scale | Assessment at baseline, after 6 weeks of intervention, 6 and 12 month post intervention
  Balance
10 meters walk test | Assessment at baseline, after 6 weeks of intervention, 6 and 12 month post intervention
  Walking
2 minutes walk test | Assessment at baseline, after 6 weeks of intervention, 6 and 12 month post intervention
  Walking
Functional Ambulation Categories | Assessment at baseline, after 6 weeks of intervention, 6 and 12 month post intervention
  Walking
Borg Rating of Perceived Exertion Scale (RPE) | Assessment at baseline, after 6 weeks of intervention, 6 and 12 month post intervention
  Interview
Montreal Cognitive Assessment | Assessment at baseline, after 6 weeks of intervention, 6 and 12 month post intervention
Hospital anxiety and Depression Scale | Assessment at baseline, after 6 weeks of intervention, 6 and 12 month post intervention
  Interview
Barthel Index | Assessment at baseline, after 6 weeks of intervention, 6 and 12 month post intervention
  Independence in mobility and personal care
Stroke Impact Scale | Assessment at baseline, after 6 weeks of intervention, 6 and 12 month post intervention
  Functioning and disability, Interview
Physical activity in everyday life using SenseWear | Assessment at baseline, after 3 weeks of intervention, after 6 weeks of intervention, 6 and 12 month post intervention
  Registers physical activity in everyday life
Objectively quantify the impairment caused by a stroke, using the National Institutes of Health Stroke Scale (NIHSS) | Assessment at baseline
  Stroke severity
Modified Ranking Scale | Assessment at baseline
  Interview
Body Mass Index | Assessment at baseline, after 6 weeks of intervention, 6 and 12 month post intervention
Weight | Assessment at baseline, after 6 weeks of intervention, 6 and 12 month post intervention
Height | Assessment at baseline, after 6 weeks of intervention, 6 and 12 month post intervention
Blood pressure | Assessment at baseline, after 6 weeks of intervention, 6 and 12 month post intervention
  Registered in everyday life
HbA1c | Assessment at baseline, after 6 weeks of intervention, 6 and 12 month post intervention
  Blood test
Plasma lipid profile | Assessment at baseline, after 6 weeks of intervention, 6 and 12 month post intervention
  Blood test
Perception of the intervention | after 6 weeks of intervention
  Interview. Study group using Hybrid Assistive Limb (HAL) only.
Smoking | Assessment at baseline, after 6 weeks of intervention, 6 and 12 month post intervention
  Interview
Alcohol | Assessment at baseline, after 6 weeks of intervention, 6 and 12 month post intervention
  Interview
Drug use | Assessment at baseline, after 6 weeks of intervention, 6 and 12 month post intervention
  From medical records
Health care consumption | 12 month post intervention
  From County Council
Stroke type and localization | At baseline
  From medical records
Dysexecutive Questionnaire | At baseline
  Filled in by significant other

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation Medicine, Danderyd Hospital, Danderyd, Stockholm County, Sweden

REFERENCES:
- [Background] Nilsson A, Vreede KS, Haglund V, Kawamoto H, Sankai Y, Borg J. Gait training early after stroke with a new exoskeleton--the hybrid assistive limb: a study of safety and feasibility. J Neuroeng Rehabil. 2014 Jun 2;11:92. doi: 10.1186/1743-0003-11-92. PMID 24890413
- [Background] Wall A, Borg J, Palmcrantz S. Clinical application of the Hybrid Assistive Limb (HAL) for gait training-a systematic review. Front Syst Neurosci. 2015 Mar 25;9:48. doi: 10.3389/fnsys.2015.00048. eCollection 2015. PMID 25859191
- [Derived] Bergqvist M, Moller MC, Bjorklund M, Borg J, Palmcrantz S. The impact of visuospatial and executive function on activity performance and outcome after robotic or conventional gait training, long-term after stroke-as part of a randomized controlled trial. PLoS One. 2023 Mar 9;18(3):e0281212. doi: 10.1371/journal.pone.0281212. eCollection 2023. PMID 36893079
- [Derived] Palmcrantz S, Wall A, Vreede KS, Lindberg P, Danielsson A, Sunnerhagen KS, Hager CK, Borg J. Impact of Intensive Gait Training With and Without Electromechanical Assistance in the Chronic Phase After Stroke-A Multi-Arm Randomized Controlled Trial With a 6 and 12 Months Follow Up. Front Neurosci. 2021 Apr 22;15:660726. doi: 10.3389/fnins.2021.660726. eCollection 2021. PMID 33967683